CLINICAL TRIAL: NCT00181714
Title: Prevention of Cigarette Smoking in ADHD Youth With Concerta
Brief Title: Prevention of Cigarette Smoking in Attention Deficit Hyperactivity Disorder (ADHD) Youth With Concerta
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief, Clinical and Research Programs in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2003-P-001313
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2012-02-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: ADHD
Keywords: cigarette smoking; ADHD; adolescents; Concerta
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Cigarette Smoking | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OROS MPH (Experimental): Single arm- open treatment with extended duration methylphenidate (OROS MPH)
  Interventions: Drug: methylphenidate HCl (Concerta)

INTERVENTIONS:
Drug: methylphenidate HCl (Concerta) — OROS MPH will be openly prescribed to a maximum of 1.5 mg/kg/day (maximum 126 mg/day). Doses will be titrated according to clinical assessment of efficacy and tolerability.
  Other Names: Concerta

SUMMARY:
This study will consist of a six-week open-label treatment period with an extended duration methylphenidate (OROS MPH) followed by subsequent monthly visits for 24 months in a large sample of youths aged 12-17 who meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for ADHD.

The researchers hypothesize that OROS MPH treatment will be associated with low rates of cigarette smoking in ADHD youth.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent outpatients between 12 to 17 years of age (inclusive).
2. Subjects with the DSM-IV diagnosis of ADHD, as manifested in the clinical evaluation and confirmed by structured interview.
3. Subjects with sufficient current ADHD symptoms to warrant treatment, as measured by a Clinical Global Impression Severity Scale (CGI-S) score of greater than or equal to 4 (moderately ill); OR subjects already on Concerta who are judged to be responders (CGI of 1 or 2) and who tolerate treatment well.

Exclusion Criteria:

1. Any serious or unstable medical illness including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease, hypertension), endocrinologic, neurologic, immunologic, or hematologic disease.
2. Clinically significant abnormal baseline laboratory values
3. History of seizures
4. Active tic disorder
5. Pregnant or nursing females
6. Mental retardation (intelligence quotient [IQ] < 75)
7. Organic brain disorder
8. Eating disorders
9. Psychosis
10. Current bipolar disorder (current episode)
11. Current depression > mild (CGI-S > 3)
12. Current anxiety > mild (CGI-S > 3)
13. Substance abuse or dependence within the past 2 months
14. Recent change in non-monoamine oxidase inhibitor (MAOI) antidepressants (< 3 months)
15. Recent change in benzodiazepines (< 3 months)
16. Concerta non-responder

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2003-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Hammerness P, Fried R, Petty C, Meller B, Biederman J. Assessment of cognitive domains during treatment with OROS methylphenidate in adolescents with ADHD. Child Neuropsychol. 2014;20(3):319-27. doi: 10.1080/09297049.2013.790359. Epub 2013 May 2. PMID 23639146
- [Derived] Hammerness P, Biederman J, Petty C, Henin A, Moore CM. Brain biochemical effects of methylphenidate treatment using proton magnetic spectroscopy in youth with attention-deficit hyperactivity disorder: a controlled pilot study. CNS Neurosci Ther. 2012 Jan;18(1):34-40. doi: 10.1111/j.1755-5949.2010.00226.x. Epub 2010 Dec 8. PMID 21143432
- [Derived] Hammerness P, Wilens T, Mick E, Spencer T, Doyle R, McCreary M, Becker J, Biederman J. Cardiovascular effects of longer-term, high-dose OROS methylphenidate in adolescents with attention deficit hyperactivity disorder. J Pediatr. 2009 Jul;155(1):84-9, 89.e1. doi: 10.1016/j.jpeds.2009.02.008. Epub 2009 Apr 25. PMID 19394037

RESULTS

PARTICIPANT FLOW:
Groups:
- OROS-Methylphenidate: Youth ages 12-17 years with DSM-IV ADHD, treated with open-label OROS-MPH.
Period: Signed Consent/Enrolled
Arm/Group | OROS-Methylphenidate
Started | 203
Completed | 154
Not Completed | 49
Period: Began Treatment With OROS-MPH
Arm/Group | OROS-Methylphenidate
Started | 154
Completed | 30
Not Completed | 124

BASELINE CHARACTERISTICS:
Arm/Group | OROS-Methylphenidate
Number analyzed (Participants) | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 154
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 114
Region of Enrollment [Number; unit: participants]
  United States | 154

OUTCOME MEASURES:

1. Primary Outcome: Cigarette Smoking
Description: Cigarette smoking was assessed by youth self report using a modified version of the Fagerstrom Tolerance Questionnaire (FTQ)
Time Frame: 24 months
Population: Clinical trial subjects included in this analysis included those adolescents who took at least one dose of OROS MPH following baseline assessment (N=154), with the last observation carried forward (LOCF) for subjects who did not complete the full study schedule of 24 months
Measure: Number; unit: percent
Arm/Group | OROS-Methylphenidate
Number analyzed (Participants) | 154
percent | 7

ADVERSE EVENTS:
Arm/Group | OROS-Methylphenidate
Serious Adverse Events (participants affected / at risk) | 5/154
Other Adverse Events (participants affected / at risk) | 45/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OROS-Methylphenidate (N=154)
leg fracture (Injury, poisoning and procedural complications) | 2 (2)
viral illness (General disorders) | 1 (2)
spontaneous pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
unintentional carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.001% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OROS-Methylphenidate (N=154)
TMJ (Musculoskeletal and connective tissue disorders) | 1 (1)
acne (Skin and subcutaneous tissue disorders) | 4 (8)
allergies (General disorders) | 3 (4)
anxiety (Psychiatric disorders) | 2 (2)
asthma attack (Respiratory, thoracic and mediastinal disorders) | 1 (1)
back pain (General disorders) | 1 (1)
jumbled thoughts (General disorders) | 1 (1)
chest pain (General disorders) | 2 (3)
cold symptoms (General disorders) | 2 (3)
congestion (General disorders) | 4 (4)
costosternal muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
cranky (General disorders) | 2 (3)
decreased appetite (General disorders) | 19 (27)
decreased energy (General disorders) | 3 (3)
deer tick bite (Injury, poisoning and procedural complications) | 1 (1)
dental infection (Infections and infestations) | 1 (2)
diarrhea (Gastrointestinal disorders) | 3 (3)
dizziness (General disorders) | 4 (5)
dull (General disorders) | 1 (1)
ear pain (Ear and labyrinth disorders) | 3 (3)
foot pain (General disorders) | 2 (2)
hand lesion (Injury, poisoning and procedural complications) | 1 (1)
headache (General disorders) | 14 (25)
heart racing (General disorders) | 6 (8)
hoarse voice (General disorders) | 1 (1)
hot/cold flashes (General disorders) | 1 (1)
hyper (General disorders) | 1 (1)
increased urination (Renal and urinary disorders) | 1 (1)
infected ingrown tonail (Infections and infestations) | 1 (1)
inflamed adenoids (General disorders) | 1 (2)
initial insomnia (General disorders) | 4 (6)
insomnia (General disorders) | 7 (8)
irritable (General disorders) | 3 (4)
jittery (General disorders) | 2 (3)
knee pain (General disorders) | 1 (2)
lightheadedness (General disorders) | 2 (2)
low interest (General disorders) | 1 (1)
menstrual cramps (Reproductive system and breast disorders) | 1 (2)
moody (General disorders) | 2 (2)
muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 4 (4)
nose bleed (General disorders) | 1 (1)
orthodontic pain (General disorders) | 1 (2)
otitis (General disorders) | 1 (1)
pain extension in bilateral arms/legs (Musculoskeletal and connective tissue disorders) | 1 (1)
phinorhea (General disorders) | 1 (1)
rapid pulse (General disorders) | 1 (5)
rash (poison ivy) (Skin and subcutaneous tissue disorders) | 1 (1)
runny nose (General disorders) | 2 (2)
sad (General disorders) | 1 (1)
shoulder pain (General disorders) | 1 (1)
sore throat (General disorders) | 4 (4)
stomach ache (Gastrointestinal disorders) | 2 (2)
teary (General disorders) | 1 (1)
tense (General disorders) | 1 (1)
tight breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
toothache (General disorders) | 1 (1)
twisted ankle pain (General disorders) | 1 (1)
upper respiratory infection (Infections and infestations) | 5 (8)
vomiting (Gastrointestinal disorders) | 2 (2)
weight loss (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The main limitation of this report stems from its uncontrolled, open-label design. Thus, we cannot assert a causal relationship between lower smoking rates and OROS MPH prescription.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes